CLINICAL TRIAL: NCT00635739
Title: Efficacy of Whey Protein Supplementation on Resistance Exercise-Induced Changes in Muscle Strength, Fat Free Mass, and Function in Mobility-Limited Older Adults
Brief Title: Effect of Whey Protein Supplementation and Resistance Exercise on Muscle Parameters in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Principal Investigator, Roger A Fielding, Director and Senior Scientist, Professor of Nutrition, Jean Mayer USDA Human Nutrition Research Center on Aging., Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1493
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-12

CONDITIONS: Mobility Limitation
Keywords: Whey protein; Resistance exercise; Physical activity; Mobility disability; Physical function; Muscle mass; Muscle strength; Older Adults; Mobility-Limited
MeSH Terms: conditions — Mobility Limitation; Motor Activity | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, 1 (Active Comparator)
  Interventions: Dietary Supplement: Whey protein
- A, 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin placebo

INTERVENTIONS:
Dietary Supplement: Whey protein — powdered, 46g supplement dissolved in fluids, twice daily
  Arms: A, 1
Dietary Supplement: Maltodextrin placebo — powdered, 46g supplement dissolved in fluids, twice daily
  Arms: A, 2

SUMMARY:
This research study is looking at the effects of a whey protein nutritional supplement on changes in muscle mass, strength and physical function in response to a 6 month program of strength training exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male and Females 70-85 yrs
* Community dwelling
* Short Physical Performance Battery score < 10
* BMI = 21-32.5

Exclusion Criteria:

* Acute or terminal illness
* Mini Mental State Exam < 23
* Myocardial infarction in previous 6 months, symptomatic coronary artery disease, or congestive heart failure
* Upper or lower extremity fracture in previous 6 months
* Uncontrolled hypertension (>150/90 mm Hg).
* Neuromuscular diseases and drugs which affect neuromuscular function.
* Hormone replacement therapy
* eGFR <30 mL/min/1.73m2
* Types I and II Diabetes Mellitus
* Dietary protein intake < 0.8 g.kg-1.day-1
* Disorders of nutrient absorption
* Milk, or whey allergy
* Sulfa drugs and allergy to PABA-containing sunscreens

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Fielding, Ph.D., Principal Investigator — Jean Mayer USDA Human Nutrition Research Center on Aging
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chale A, Cloutier GJ, Hau C, Phillips EM, Dallal GE, Fielding RA. Efficacy of whey protein supplementation on resistance exercise-induced changes in lean mass, muscle strength, and physical function in mobility-limited older adults. J Gerontol A Biol Sci Med Sci. 2013 Jun;68(6):682-90. doi: 10.1093/gerona/gls221. Epub 2012 Oct 31. PMID 23114462

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Maltodextrin placebo: powdered, 46g supplement dissolved in fluids, twice daily
Period: Overall Study
Arm/Group | Whey Protein | Placebo
Started | 42 | 38
Completed | 39 | 36
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- A,1 (Intervention): Whey protein: powdered, 46g supplement dissolved in fluids, twice daily
- A,2 (Control): Maltodextrin placebo: powdered, 46g supplement dissolved in fluids, twice daily
- Total: Total of all reporting groups
Arm/Group | A,1 (Intervention) | A,2 (Control) | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (4.0) | 77.3 (3.9) | 77.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 42 | 38 | 80

OUTCOME MEASURES:

1. Primary Outcome: 1 Repetition Maximum Muscle Strength 1-RM (N) Double Leg Press
Description: The maximum muscle strength of the leg extensor muscles as measured by pneumatic strength training equipment.
Time Frame: Baseline and follow up (6 months)
Population: 5 subjects were not included in follow up analysis
Measure: Mean (Standard Deviation); unit: N
Arm/Group | Whey Protein | Placebo
Number analyzed (Participants) | 42 | 38
N
  Baseline | 1223 (380) | 1256 (461)
  Follow up: number analyzed (Participants) | 39 | 36
  Follow up | 1483 (517) | 1465 (528)

2. Secondary Outcome: Lean Mass
Description: Whole body lean mass (kg) as measured by dual energy x-ray absorptiometry.
Time Frame: Baseline and follow up (6 months)
Population: 5 subjects were not included in follow up analysis
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Whey Protein | Placebo
Number analyzed (Participants) | 42 | 38
Kg
  Baseline | 46.7 (8.6) | 46.4 (8.4)
  Follow up: number analyzed (Participants) | 39 | 36
  Follow up | 47.3 (8.6) | 46.7 (8.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Whey Protein | Placebo
Serious Adverse Events (participants affected / at risk) | 6/42 | 3/38
Other Adverse Events (participants affected / at risk) | 14/42 | 19/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Whey Protein (N=42) | Placebo (N=38)
Cardiovascular (Cardiac disorders) | 2 | 1
fall (General disorders) | 1 | 1
hospitalization (General disorders) | 3 | 1 — Hospitalization reason is not know.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whey Protein (N=42) | Placebo (N=38)
GI distress (Gastrointestinal disorders) | 4 (4) | 2 (2) — GI upset
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Non-injurious fall
Surgery (Surgical and medical procedures) | 1 (1) | 5 (5) — Outpatient surgical procedure
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) — Musculoskeletal pain/injury
Laboratory (General disorders) | 3 (3) | 1 (1) — Abnormal laboratory value
Illness (General disorders) | 5 (5) | 6 (6) — Illness that would restrict physical activity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No